CLINICAL TRIAL: NCT04465916
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Study of Oral FXR Modulator EYP001a Combined With Nucleos(t)Ide Analogues (NA) in Virologically Suppressed Chronic Hepatitis B Patients to Improve Functional Cure Rates
Brief Title: Study of EYP001a to Assess Its Safety and Anti-viral Effect in CHB Patients in Combination With NA (ETV or TD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMC reviewed results of 26 subjects. New randomizations were stopped. Already randomized subjects were followed up to W40.
Sponsor: Enyo Pharma (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry); Synteract, Inc. (Industry); Eurofins (Industry); Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EYP001-201
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Experimental Arm: EYP001a Dose A QD + NA daily (37 patients)
  Interventions: Drug: EYP001a; Drug: Nucleotide analogue (Entecavir or Tenofovir Disoproxil)
- Control Arm (Placebo Comparator): Control Arm: Placebo + NA daily (12 patients)
  Interventions: Drug: Placebo; Drug: Nucleotide analogue (Entecavir or Tenofovir Disoproxil)

INTERVENTIONS:
Drug: EYP001a — Oral tablets
  Arms: Experimental Arm
Drug: Placebo — Oral tablets
  Arms: Control Arm
Drug: Nucleotide analogue (Entecavir or Tenofovir Disoproxil) — Oral tablets

SUMMARY:
This is a prospective, multi-centre, randomized, double-blind, placebo-controlled, Phase 2a experimental study of oral FXR modulator EYP001a/placebo combined with NAs in virologically suppressed CHB patients to improve functional cure rates.

DETAILED DESCRIPTION:
A total of 49 eligible patients will be enrolled and randomized at approximately 14 study sites. Patients will be randomized prior to study drug (EYP001a or placebo and NA) administration on Day 1 in the ratio of 3:1 into 2 arms:

* Experimental Arm: EYP001a Dose A QD + NA daily (37 patients)
* Control Arm: Placebo + NA daily (12 patients)

The maximum total engagement duration for eligible patients in this study is up to 370 days: 90 days screening, 112 days (16 weeks) treatment period and 168 days (24 weeks) follow-up.

Patients enrolled in the study will be assessed as outpatients. Patient screening will occur no more than 90 days prior to the Day 1 visit. Eligible patients will undergo further assessments on Day 1 to qualify for study drug administration on Day 1.

The visits during the study are planned as below:

* Screening visit: 12 weeks (90 days)
* 16 weeks treatment period:
* Treatment Visit 1 (Week 1 [Day 1])
* Treatment Visit 2 (Week 2 [Day 14 ±3 days])
* Treatment Visit 3 (Week 4 [Day 28 ±3 days])
* Treatment Visit 4 (Week 6 [Day 42 ±3 days])
* Treatment Visit 5 (Week 8 [Day 56 ±3 days])
* Treatment Visit 6 (Week 10 [Day 70 ± 3 days])
* Treatment Visit 7 (Week 12 [Day 84 ± 3 days])
* Treatment Visit 8 (Week 14 [Day 98 ± 3 days])
* Treatment Visit 9 (Week 16 [Day 112±3 days])
* 24 weeks safety follow-up period:
* Follow-up Visit 1 (Week 20 [Day 140 ±7 days])
* Follow-up Visit 2 (Week 28 [Day 196 ±7 days])
* Follow-up Visit 3 (Week 40 [Day 280 ±7 days]) Note: during follow-up patients are kept on NA until the end of the trial: Week 40 (consolidation Phase).

ELIGIBILITY:
Main Inclusion Criteria:

* Are on stable NA therapy at least 12 months from the screening date (ETV or TDF)
* Has virally suppressed CHB:

HBV DNA <LLOQ and serum HBsAg >100 IU/mL

* Has liver imaging to screen for hepatocellular carcinoma or concomitant pancreaticobiliary disease either in the prior 6 months or at screening.
* Is not of childbearing potential or, if of childbearing potential, is not pregnant as confirmed by a negative serum human chorionic gonadotropin test at screening and is not planning a pregnancy during the course of the study.

Main Exclusion Criteria:

* Is an employee of a contract research organization (CRO), vendor, or Sponsor involved with this study.
* Has known hepatocellular carcinoma or pancreaticobiliary disease.
* Neutropenia (defined by two confirmed values within screening period of <1500/μL).
* Has Gilbert syndrome.
* Shows evidence of worsening liver function, defined as either a confirmed (two assessments at least 3 days apart) increase >2 ULN ALT or AST or an increase of >1.5 × first assessed value of TBL or associated with clinical signs or symptoms of liver impairment.
* Has known or suspected non-CHB liver disease
* History of cirrhosis or liver decompensation, including ascites, hepatic encephalopathy, or presence of oesophageal varices.
* Probable or possible F3 stage with a vibration controlled transient elastography (VCTE). Patients with normal baseline ALT and VCTE >8.8 kPa are excluded. Patients with baseline ALT >ULN (but <2ULN per EC5) and who have VCTE >10.5 kPa at baseline are excluded 11.
* Has known history of alcohol abuse or daily heavy alcohol consumption
* Has clinically relevant immunosuppression, including, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
* Has used anti-HBV medications other than NAs within 90 days prior to screening.
* Has any of the following exclusionary laboratory results at screening:

  1. Estimated glomerular filtration rate <60 mL/min/1.73 m2 (the Modification of Diet in Renal Disease formula).
  2. Thyroid-stimulating hormone >1.5× ULN or abnormal free triiodothyronine or free thyroxine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ENYO PHARMA Investigative site KR04, Principal Investigator — Pusan, South Korea; ENYO PHARMA Investigative site KR03, Principal Investigator — Seoul, South Korea; ENYO PHARMA Investigative site KR02, Principal Investigator — Seoul, South Korea; ENYO PHARMA Investigative site KR01, Principal Investigator — Seoul, South Korea; ENYO PHARMA Investigative site PL06, Principal Investigator — Kielce, Poland; ENYO PHARMA Investigative site PL05, Principal Investigator — Łódź, Poland; ENYO PHARMA Investigative site PL04, Principal Investigator — Zawiercie, Poland; ENYO PHARMA Investigative site PL03, Principal Investigator — Warszawa, Poland; ENYO PHARMA Investigative site PL02, Principal Investigator — Lublin, Poland; ENYO PHARMA Investigative site PL01, Principal Investigator — Białystok, Poland; ENYO PHARMA Investigative site AU04, Principal Investigator — Melbourne, Australia; ENYO PHARMA Investigative site AU03, Principal Investigator — Melbourne, Australia; ENYO PHARMA Investigative site AU02, Principal Investigator — Brisbane, Australia; ENYO PHARMA Investigative site AU01, Principal Investigator — Melbourne, Australia; ENYO PHARMA Investigative site HK01, Principal Investigator — Hong Kong, Hong Kong; ENYO PHARMA Investigative site KR05, Principal Investigator — Seongnam, South Korea; ENYO PHARMA Investigative site KR06, Principal Investigator — Séoul, South Korea; ENYO PHARMA Investigative site KR07, Principal Investigator — Pusan, South Korea
Locations (18):
- Australia (4):
  - ENYO PHARMA Investigative site AU02, Brisbane
  - ENYO PHARMA Investigative site AU01, Melbourne
  - ENYO PHARMA Investigative site AU03, Melbourne
  - ENYO PHARMA Investigative site AU04, Melbourne
- ENYO PHARMA Investigative site HK01, Hong Kong, Hong Kong
- Poland (6):
  - ENYO PHARMA Investigative site PL01, Bialystok
  - ENYO PHARMA Investigative site PL06, Kielce
  - ENYO PHARMA Investigative site PL05, Lodz
  - ENYO PHARMA Investigative site PL02, Lublin
  - ENYO PHARMA Investigative site PL03, Warsaw
  - ENYO PHARMA Investigative site PL04, Zawiercie
- South Korea (7):
  - ENYO PHARMA Investigative site KR04, Pusan
  - ENYO PHARMA Investigative site KR07, Pusan
  - ENYO PHARMA Investigative site KR05, Seongnam
  - ENYO PHARMA Investigative site KR01, Seoul
  - ENYO PHARMA Investigative site KR02, Seoul
  - ENYO PHARMA Investigative site KR03, Seoul
  - ENYO PHARMA Investigative site KR06, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Experimental Arm: EYP001a 200 mg daily + Nucleotide analogue daily (37 patients)
  EYP001a: Oral tablets
  Nucleotide analogue (Entecavir or Tenofovir Disoproxil): Oral tablets
- Control Arm: Control Arm: Placebo daily + Nucleotide analogue daily (12 patients)
  Placebo: Oral tablets
  Nucleotide analogue (Entecavir or Tenofovir Disoproxil): Oral tablets
Period: Overall Study
Arm/Group | Experimental Arm | Control Arm
Started | 19 | 7
Completed | 19 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Control Arm | Total
Number analyzed (Participants) | 19 | 7 | 26
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 45.16 (8.32) | 46.29 (8.46) | 45.46 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 14 | 6 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 19 | 5 | 24
  Black or African American | 0 | 1 | 1
  White | 0 | 1 | 1
Weight [Geometric Mean (Standard Deviation); unit: kg] | 68.821 (11.293) | 82.857 (21.084) | 72.600 (15.454)
Height [Geometric Mean (Standard Deviation); unit: cm] | 168.763 (9.333) | 172.529 (11.342) | 169.777 (9.823)

OUTCOME MEASURES:

1. Primary Outcome: HBsAg Change (Δ log10) From Day 1 to Week 16 of Treatment
Description: Efficacy of Vonafexor on top of NA assessed as HBsAg decline (Δ log10) from Day 1 to Week 16 of treatment
Time Frame: LS mean at week 16 (Day 1, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 14, and Week 16)
Measure: Least Squares Mean (Standard Error); unit: log10 IU/mL
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 19 | 7
log10 IU/mL | -0.029 (0.0195) | -0.066 (0.0348)

2. Secondary Outcome: Virologic Failure Rate
Description: Virologic failure rate (breakthrough)2 of HBV-DNA (% patients with a confirmed quantifiable HBV DNA increase of ≥ 1log10 HBV DNA copies/mL above LLOQ3) assessed at Week 16 of treatment period and Weeks 20, 28 and 40 during follow-up period
Time Frame: 40 weeks
Measure: Number; unit: participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 19 | 6
participants
  Week 16 | 0 | 0
  Week 20 | 0 | 0
  Week 28 | 0 | 0
  Week 40 | 0 | 0

ADVERSE EVENTS:
Time Frame: After the first dose of study drug until W40
Description: Participants received either Entecavir or Tenofovir Disoproxil Fumarate in each Arm/Group combined with Placebo or EYP001.
  Entecavir and Tenofovir Disoproxil Fumarate are both NA and are therapeutically equivalent.
  Therefore safety results are presented for Experimental Arm and Control Arm irrespective of NA therapy taken.
Arm/Group | Experimental Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/7
Other Adverse Events (participants affected / at risk) | 17/19 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=19) | Control Arm (N=7)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Vaccination site discomfort (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (19) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data may be considered for publication in a scientific journal or for reporting at a scientific meeting. Each Investigator is obligated to keep data pertaining to the study confidential. The Investigator must consult with the Sponsor before any study data are submitted for publication. The Sponsor reserves the right to deny publication rights until mutual agreement on the content, format, interpretation of data in the manuscript, and journal selected for publication are achieved.

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04465916/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT04465916/SAP_001.pdf